CLINICAL TRIAL: NCT01083485
Title: A Randomised, Double-blind, Parallel Group Multicentre Study to Demonstrate Non-inferiority of the Analgesic Efficacy of Oxycodone/Naloxone 10/5 or 20/10 mg Prolonged Release Tablets (OXN PR) BID Compared to Oxycodone 10 or 20 mg Prolonged Release Tablets (OXY PR) BID in Subjects With Postoperative Pain After Knee Arthroplasty
Brief Title: OXN PR Compared to OXY PR in Subjects With Postoperative Pain After Knee Arthroplasty
Acronym: OXN4505
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXN4505; 2009-016957-17 (EudraCT Number)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Results first posted 2012-02-16 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Post Operative Pain
Keywords: Oxycodone; Naloxone; Postoperative pain; Arthroplasty; Efficacy
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablets Oxycodone Naloxone (OXN) (Experimental): Oxycodone/Naloxone prolonged release 20/10mg or 10/5mg tabs twice a day (BID) for 2.5 days (total 5 dosages)
  Interventions: Drug: Oxycodone/Naloxone PR 20/10mg or 10/5mg tablets
- Oxycodone (Active Comparator): Oxycodone PR 20mg or 10mg (twice a day) BID for 2.5 days (total 5 dosages)
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone/Naloxone PR 20/10mg or 10/5mg tablets — Oxycodone/Naloxone prolonged release 20/10mg or 10/5mg tabs twice a day (BID) for 2.5 days (total 5 dosages)or Oxycodone 20mg
  Arms: Tablets Oxycodone Naloxone (OXN)
Drug: Oxycodone — Oxycodone 20mg or 10mg BID for 2.5 days (total 5 dosages)
  Arms: Oxycodone

SUMMARY:
The purpose of this study is to demonstrate that treatment with OXN PR tablets is non inferior to treatment with OXY PR tablets in terms of analgesic efficacy in patients with postoperative pain after knee arthroplasty based on average pain intensity scores.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 - 75 years of age.
* Body mass index (BMI) 18 - 35 kg/m2.
* If female and less than one year post-menopausal:

  * negative serum or urine pregnancy test (positive beta-human chorionic gonadotrophin test) at screening.
  * using an adequate and highly effective method of contraception throughout the study. A highly effective method of contraception is defined as one with a failure rate of less than 1% per year when used consistently and correctly. Examples include sterilisation, implants, injectables, combined oral contraceptives, hormonal intra uterine devices, sexual abstinence or vasectomised partner.
* Confirmed diagnosis of osteoarthritis of the knee.
* Planned surgical arthroplasty on one knee.
* Planned postoperative epidural analgesia for approximately 48 hours.
* Anticipated requirement for daily opioid treatment after epidural analgesia for 2.5 days.
* Able to participate in the study and have given written informed consent.

Exclusion Criteria:

* Females who are pregnant or lactating.
* Opioid use within 3 months before the start of the screening period. Stable treatment with analgesics in World Health Organisation (WHO) Step I (non-opioid analgesics) is allowed.
* History of laxative use to treat constipation within 3 months before the start of the screening period.
* History of chronic constipation.
* Concurrent rheumatoid arthritis.
* Planned bilateral arthroplasty or revision knee arthroplasty.
* History of moderate to severe hepatic impairment.
* History of moderate to severe respiratory depression with hypoxia or hypercapnia, chronic obstructive pulmonary disease, cor pulmonale, bronchial asthma, or any severe impairment of pulmonary function.
* History of uncontrolled hypothyroidism, Addison's disease (adrenal cortical insufficiency), psychosis, cholelithiasis, prostatic hypertrophy(with documented residual of over 100 ml after voiding), delirium tremens, pancreatitis, hypotension, uncontrolled hypertension, uncontrolled cardiovascular diseases, head injury, epileptic disorder or predisposition to convulsions, or treatment with monoamine oxidase inhibitors (concurrent or within 2 weeks of discontinuation).
* Contraindication to treatment with opioids.
* History of hypersensitivity to oxycodone, naloxone, or to any of the excipients of OXN PR tablets.
* History of non-opioid induced paralytic ileus.
* Previous or current history of drug abuse, including alcohol abuse or opioid abuse.
* Evidence of clinically unstable disease
* Receipt of an investigational medicinal product within 30 days before the start of the screening period.
* Galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* Delayed gastric emptying.
* Severe renal impairment (i.e. creatinine clearance <10 mL/minute).
* Weight <50 kg.Inclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Central hospital of Pori, Pori, Finland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit 25 March 2010 and last patient last visit 17 Oct 2010. Five Hospital Investigator Centres
Pre-assignment Details: 14 day screening period before planned surgery. Run-in period 48 hours, 2.5 day double-blind period after surgery
Groups:
- OXN Tablets: Oxycodone/Naloxone prolonged release (PR) 20/10mg or 10/5mg tablets twice a day (BID) for 2.5 days (total = 5 doses)
- OXY Tablets: Oxycodone prolonged release (PR) 20mg or 10mg tablets twice a day (BID) for 2.5 days (total = 5 doses)
Period: Overall Study
Arm/Group | OXN Tablets | OXY Tablets
Started | 70 | 67
Completed | 63 | 64
Not Completed | 7 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OXN Tablets | OXY Tablets | Total
Number analyzed (Participants) | 70 | 67 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 33 | 69
  >=65 years | 34 | 34 | 68
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (6.7) | 64 (6.7) | 64 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 39 | 83
  Male | 26 | 28 | 54
Region of Enrollment [Number; unit: participants]
  Finland | 70 | 67 | 137

OUTCOME MEASURES:

1. Primary Outcome: Mean of 4 NRS Scores for 24 Hour Pain Intensity at Rest, Shown as Absolute Change From Baseline (i.e. a Decrease From the Baseline Value)
Description: The primary efficacy variable was the 24hr pain intensity score at rest, on a Numerical Rating Scale (NRS), with "0" = "no pain" and "10" = "worst possible pain". This was assessed 1 hour after dosing on Day 1 (evening only), Day 2(morning and evening) and Day 3 (morning only). The primary efficacy end point (absolute change from baseline) was analysed on the per protocol (PP) data. The mean of these scores is shown as a value that is a mean change (a decrease in pain score) from the baseline value.
Time Frame: Mean of 24 hour pain intensity (absolute change from baseline)
Population: The primary efficacy end point (absolute change from baseline) was analysed on the PP data using a mixed model repeated measures of analysis of covariance (RMANCOVA).
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- OXN Tablets: Oxycodone/Naloxone prolonged release (PR) 20/10mg or 10/5mg tablets twice a day (BID) for 2.5 days (total = 5 doses). Mean baseline pain score = 3.4
- OXY Tablets: Oxycodone prolonged release (PR) 20mg or 10mg tablets twice a day (BID) for 2.5 days (total = 5 doses). Mean baseline pain score = 3.1
Arm/Group | OXN Tablets | OXY Tablets
Number analyzed (Participants) | 59 | 62
Units on a scale | -1.2 [-1.5 to -0.9] | -1.1 [-1.4 to -0.8]
Statistical Analysis 1: Comparison: OXN Tablets vs OXY Tablets; The sample size was calculated for a significance level of 2.5% (1 sided) with 90% power. A within SD 1.7, and expected treatment difference of 0 and a non-inferiority margin of 1.0 were assumed; Test type: Non-Inferiority or Equivalence — Previously provided; ANCOVA — A P value was not part of the analysis plan. A within SD 1.7, and expected treatment difference of 0 and a non-inferiority margin was -1.0 meaning that OXN PR can be one unit inferior to OXY PR and still be considered non-inferior; The primary efficacy endpoint was analysed on the PP data using a mixed-model repeat measure analysis of covariance RMANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.5 to 0.3]

2. Secondary Outcome: Mean Dose (mg) of Rescue Analgesia for the Treatment Phase for Subjects Taking 20/10mg OXN PR Tablets or 20mg OXY PR Tablets
Description: To compare the use of rescue analgesia for the 2 groups (OXN 20/10mg tablets and OXY 20mg tablets) during the double blind treatment phase. Rescue medication was given (OXY Immediate Release, 5mg capsules) if the subjects pain score on the (Numeric Rating Scale (NRS), 0 (no pain) to 10 (worst possible pain)), was greater than or equal to 4. The value presented is the mean dose over the double blind phase.
Time Frame: Mean dose during the whole double blind treatment phase (2.5 days)
Population: This is the per protocol population (PP), which is a subset of the full analysis population. The data presented is only for those subjects taking the higher dose (20/10 mg OXN or 20 mg OXY) in the study.
Measure: Mean (Standard Deviation); unit: mg of rescue analgesia
Arm/Group | OXN Tablets | OXY Tablets
Number analyzed (Participants) | 36 | 33
mg of rescue analgesia | 24 (28.7) [3.8 to 9.3] | 17 (25.4) [5.9 to 18.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from informed consent until participation in trial was completed, this could be a minimum of 1 day to a maximum of 23 days.
Description: Adverse events were collected by spontaneous question and causality and severity were assigned by the investigator.
Arm/Group | OXN Tablets | OXY Tablets
Serious Adverse Events (participants affected / at risk) | 2/70 | 0/67
Other Adverse Events (participants affected / at risk) | 43/70 | 39/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OXN Tablets (N=70) | OXY Tablets (N=67)
Mild pyrexia (General disorders) | 1 (1) | 0 (0)
severe neuropathic pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OXN Tablets (N=70) | OXY Tablets (N=67)
abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 26 (26) | 22 (22)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 7 (7) | 8 (8)
vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
chest pain (General disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
pain (General disorders) | 0 (0) | 1 (1)
pyrexia (General disorders) | 0 (0) | 2 (2)
excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 3 (3) | 0 (0)
confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
hallucination visual (Psychiatric disorders) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No